CLINICAL TRIAL: NCT02894762
Title: Performance Evaluation of In-Vitro Diagnostic Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lite-On Technology Corporation H.S.P.B (Industry)
Responsible Party: Sponsor
Other Study IDs: 201410068DSD
Record Dates: First submitted 2016-08-16; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Blood Routine Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This is an interim report for POC testing of skyla Clinical Chemistry Analyzer and four skyla Test Systems (ALB, BUN, GLU, and TP). The analyses are performed with skyla Clinical Chemistry Analyzer.

Analyte Principle:

Albumin (ALB) - Dye-Binding BCG

Blood urea nitrogen (BUN) - Urease with GLDH (coupled enzyme)

Glucose (GLU) - Hexokinase, Colorimetry

Total Protein (TP) - Biuret

ELIGIBILITY:
Inclusion Criteria:

* You must be an adult over 20 years of age and weigh over 50 kg to be eligible to participate in the study.

Exclusion Criteria:

* You may not participate in this study if you do not meet the above inclusion criteria.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative measurement of biochemical indicators in the blood of adult that include of Albumin (ALB), Blood urea nitrogen (BUN), Glucose (GLU), and Total Protein (TP). | 6 months
  Measured results will collected from the at least 120 individuals of adults for each biochemical indicator.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan